CLINICAL TRIAL: NCT02888977
Title: An Observatory for Patients Aged 55 Years and Over With Philadelphia Chromosome Positive (Ph+ or BCR-ABL+) Acute Lymphoblastic Leukemia (ALL) and Treated With the Combination of Tyrosine Kinase Inhibitors and Low Intensity Chemotherapy.
Brief Title: Tyrosine Kinase Inhibitors and Low Intensity Chemotherapy in Ph+ ALL
Acronym: EWALL_OBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, Study coordinator, Versailles Hospital
Other Study IDs: 12/13_ EWALL Obs
Record Dates: First submitted 2016-08-19; First posted 2016-09-05 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Lymphoblastic Leukemia, Acute
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of imatinib in combination with chemotherapy is now considered as the gold standard for the treatment of Ph+ ALL. The complete remission (CR) rate is 90% versus 20% to 40% with chemotherapy alone. The combination of imatinib, vincristine and dexamethasone is a well tolerated regimen in aged patients and is also associated with a high CR rate of 80% to 90% in patient aged 55 years and over. 2. Dasatinib is indicated as first line therapy in Ph+ ALL. Results from the EWALLPH-01 are supporting the use of dasatinib in combination with low-intensity chemotherapy. A new EWALL-PH-02 study combining nilotinib in combination with low-intensity chemotherapy is currently initiated within the EWALL centers.

3. The EWALL-PH-01 trial is now closed after the recruitment of 71 patients. The activation of the EWALL-PH-02 trial is expected for Q1 2012. Based on the recruitment of the EWALL-PH-01 study it could be anticipated that 50 to 100 patients aged more than 55 years will be diagnosed during this 6 months period of time. In addition, all the EWALL centers are not participating to the EWALL-PH-02 study and thus these centers could be offered to treat patient following the EWALL backbone in addition to imatinib. 4. A minimum data set will be defined in order to collect the data of the patients treated following the EWALL-PH imatinib study. The main recommendation is to follow as close as possible the procedures of the EWALL-PH-01 trial (mutation analysis, MRD follow-up) in order to have a comparable data set. This imatinib treated cohort of patients would be of particular importance in order to better define the potential benefit of using one TKI compared to one other. From the end of the EWALL-PH-01 study recruitment to the initiation of the EWALL-PH-02 study, patients were treated following the common backbone schedule in combination with imatinib or others TKI. Patients not included in clinical trials for other reasons were also offered a treatment with the combination of TKIs and backbone low-intensity chemotherapy. The goal of this observatory retrospective and prospective is to describe the efficacy and the tolerance of the combination of tyrosine kinase inhibitors in combination with low intensity chemotherapy (EWALL backbone) in patients with Ph+ ALL aged 55 years and over.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 55 years
2. Philadelphia chromosome or BCR-ABL positive acute lymphoblastic leukaemia
3. Not included in a prospective clinical trial
4. Treatment with the combination of tyrosine kinase inhibitors and low dose chemotherapy as recommended by the EWALL group (EWALL backbone).

Exclusion Criteria:

1. Patients deceded and having previously refused data collection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All consecutive previously untreated patients aged 55 years and over with Philadelphia positive acute lymphoblastic leukaemia (Ph+ ALL) not included in a prospective clinical trial and treated with the combination of TKIs and low-intensity chemotherapy (EWALL backbone see Appendix 1) should be recorded in each center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The primary end-point will be Progression Free Survival (PFS) rate at 12 months | 12 months

SECONDARY OUTCOMES:
The proportion of Complete haematological remission | 12 months
The proportion of Major molecular response defined by a BCR-ABL/ABL ≤ 0.1% in bone marrow | 12 months
The proportion of Complete molecular response | 12 months
Event free survival | 12 months
Relapse free survival | 12 months
Progression free survival | 12 months
The proportion of Detection of a T315I or F317 BCR-ABL TK mutation | 12 months
The proportion of molecular progression defined by the loss of major molecular response | 12 months
Overall survival | 12 months
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rousselot philippe, MD, Principal Investigator — CH Versailles
Locations (3):
- France (3):
  - CH Versailles, Le Chesnay
  - CHU Nimes, Nîmes
  - CH Reims, Reims

IPD SHARING:
Plan to Share IPD: No